CLINICAL TRIAL: NCT04517786
Title: A Prospective, Open, Clinical Trial Analysing The Efficacy and Safety of MINIJECT (MINI SO627) In Patients With Open Angle Glaucoma Uncontrolled By Topical Hypotensive Medications Using A Single Operator Delivery Tool
Brief Title: MINIject (MINI SO627) in Patients With Open Angle Glaucoma Using Single Operator Delivery Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: iSTAR Medical (Industry)
Collaborators: International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISM10
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma, Open-Angle Glaucoma Eye
Keywords: Glaucoma; Medical device; MIGS drainage device; eye reduction IOP
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: MINIject SO627
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MINIject CS627 implant (Experimental): MINIject 627 implant is used to reduce intra-ocular pressure in the eye. It is implanted through a minimally-invasive glaucoma surgical intervention in a stand alone procedure.
  Interventions: Device: MINIject CS627 implant

INTERVENTIONS:
Device: MINIject CS627 implant — MINI SO627 is an integrated system comprising a minimally-invasive Glaucoma Drainage Implant (CS627) and a single operator delivery tool.
  The delivery tool is a single-use tool, designed for inserting the CS627 implant into the suprachoroidal space in the eye.

SUMMARY:
The study will assess safety and performance in patients with open-angle glaucoma uncontrolled by topical hypotensive medications who had previously been implanted with a MINIject glaucoma implant.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of MINI SO627 and IOP (Intra- ocular pressure) lowering effects with or without the use of glaucoma medications. The procedure will be a stand alone surgery. Patient follow up with several examinations up to 24 months after surgery.

The primary endpoint is the reduction in medicated mean diurnal IOP at 6 months follow up compared to medicated diurnal IOP at baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary open angle glaucoma during screening/baseline visit or earlier.
* Grade 3 or grade 4 according to Shaffer Angle Grading System.
* Glaucoma not adequately controlled by one to four different topical hypotensive medication(s), given each for at least one month, as confirmed by 21mmHg < IOP < 35 mmHg in the study eye at baseline visit.

Exclusion Criteria:

* Grade 2 (narrow, 20 degrees), grade 1 (extremely narrow, less or equal to 10 degrees) and grade 0 (closed or slit) according to Shaffer Angle Grading System in the study eye.
* Neovascular glaucoma in the study eye.
* Corneal opacity or iridocorneal angle not visible through gonioprism in the study eye, preventing correct placement of the implant in the stud eye.
* Prior glaucoma surgery in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in medicated or unmedicated (without washout) mean diurnal IOP at 6 months follow-up | 6 month post surgey
  The primary endpoint of the study is the reduction in medicated or unmedicated (without washout) mean diurnal IOP at 6 months follow-up compared to medicated or unmedicated (without washout) diurnal IOP at baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR
Locations (2):
- Maxivision Super Speciality Eye Hospital, Hyderabad, India
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No